CLINICAL TRIAL: NCT02759068
Title: Beneficial Effects of Preference on Behavior
Brief Title: Beneficial Effects of Preference on Behavior in DOC Patients (COGNICOMA)
Acronym: COGNICOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-882; 2014-A01062-45 (Other: ANSM)
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Disorders of Consciousness
Keywords: vegetative state; minimally conscious state; music; preference
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State | interventions — Sound; Odorants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients behavior (Experimental): Behavior (motor reaction) to stimuli (sounds and odors)
  Interventions: Behavioral: sounds and odors
- healthy volunteers behavior (Active Comparator): Behavior (motor reaction) to stimuli (sounds and odors)
  Interventions: Behavioral: sounds and odors

INTERVENTIONS:
Behavioral: sounds and odors — presentation of sounds and odors

SUMMARY:
Preferred music improves cognitive function in patients with disorders of consciousness (DOC). However, it is still unknown whether it is a general effect of music (because of its acoustic features) or an autobiographical effect (because of its emotional and meaningful contents).

The aim of the present study was to investigate the effect of sensory modality (auditory versus olfactory) and preference (preferred versus neutral) of the testing context on the performance of four items from the coma recovery scale-revised

ELIGIBILITY:
Inclusion Criteria:

* Disorders of consciousness (Traumatic brain injury, stroke or anoxic encephalopathy)
* Coma diagnosis (Plum and Posner, 1966), vegetative state (Task Force, 1994) or minimally conscious state (Giacino, Ashwal et al. 2002)
* Lack of autonomic crisis since one week minimum
* Medical condition considered stable
* Patients who do not present hearing loss. Peaks I and II of Brainstem Auditory Evoked Potentials (BAEP) will be normal.

Exclusion Criteria:

* Hearing Problem
* Uncontrolled Epilepsy
* Autonomic crises
* Medical unstable state
* Pregnant or likely to be (interrogation data) or breastfeeding woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Cognitive Function measured using the Coma Recovery Scale | within the first 30 days
  Improvement of the score following sound stimuli and/or preferred stimuli

SECONDARY OUTCOMES:
Reaction time | within the first 30 days
  Faster reaction following sound stimuli and/or preferred stimuli

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Henry Gabrielle & Hôpital Neurologique, Saint-Genis-Laval, France